CLINICAL TRIAL: NCT00072215
Title: A Randomized Phase III Study of Paclitaxel, Ifosfamide and Cisplatin Versus Vinblastine, Ifosfamide and Cisplatin as Second-Line Therapy for Patients With Relapsed/Resistant Germ Cell Tumors
Brief Title: Cisplatin and Ifosfamide Combined With Either Paclitaxel or Vinblastine in Treating Men With Progressive or Recurrent Metastatic Germ Cell Tumors
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-90106; U10CA031946 (NIH); CDR0000339340 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Extragonadal Germ Cell Tumor; Testicular Germ Cell Tumor
Keywords: recurrent malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and seminoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma; testicular embryonal carcinoma and seminoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma; testicular seminoma; testicular yolk sac tumor and teratoma with seminoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor; recurrent extragonadal non-seminomatous germ cell tumor; recurrent extragonadal seminoma; stage IV extragonadal non-seminomatous germ cell tumor; stage IV extragonadal seminoma; testicular immature teratoma; testicular mature teratoma; recurrent extragonadal germ cell tumor
MeSH Terms: conditions — Testicular Germ Cell Tumor; Testicular Neoplasms; Carcinoma, Embryonal; Seminoma; Teratoma; Endodermal Sinus Tumor | interventions — Cisplatin; Ifosfamide; Paclitaxel; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regimen A: TIP (Experimental)
  Interventions: Drug: cisplatin; Drug: ifosfamide; Drug: paclitaxel
- Regimen B: VeIP (Experimental)
  Interventions: Drug: cisplatin; Drug: ifosfamide; Drug: vinblastine

INTERVENTIONS:
Drug: cisplatin — given IV
Drug: ifosfamide — given IV
Drug: paclitaxel — given IV
  Arms: Regimen A: TIP
Drug: vinblastine — given IV
  Arms: Regimen B: VeIP

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ifosfamide, cisplatin, paclitaxel, and vinblastine, work in different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether ifosfamide and cisplatin are more effective when combined with paclitaxel or vinblastine in treating germ cell tumors.

PURPOSE: This randomized phase III trial is studying paclitaxel, ifosfamide, and cisplatin to see how well they work compared to vinblastine, ifosfamide, and cisplatin in treating men with progressive or recurrent metastatic germ cell tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival of men with progressive or recurrent metastatic germ cell tumors treated with paclitaxel, ifosfamide, and cisplatin vs vinblastine, ifosfamide, and cisplatin as second-line therapy.

Secondary

* Compare the progression-free survival of patients treated with these regimens.
* Compare the toxicity profiles of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prior complete response or partial response with negative markers for at least 6 months (yes vs no) and relapse at least 2 years after completing first-line chemotherapy for germ cell tumors (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive paclitaxel IV over 24 hours on day 1 and cisplatin IV over 20-30 minutes and ifosfamide IV over 30 minutes on days 2-5. Patients also receive filgrastim (G-CSF) subcutaneously (SC) on days 7-18 OR pegfilgrastim SC once within 24-72 hours after completion of chemotherapy.
* Arm II: Patients receive vinblastine IV on days 1 and 2 and cisplatin IV over 20-30 minutes and ifosfamide IV over 30 minutes on days 1-5. Patients also receive G-CSF SC on days 7-18 OR pegfilgrastim as in arm I.

In both arms, treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months for 2 years, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed germ cell tumor (GCT), including 1 of the following primary tumor sites:

  * Seminoma

    * Testis
    * Retroperitoneum
    * Mediastinum
    * Other extragonadal site
  * Nonseminoma

    * Testis
    * Retroperitoneum
    * Other extragonadal site

      * No tumor of the mediastinum
* Must have evidence of metastatic disease, including either of the following:

  * Unidimensionally measurable lesions

    * At least 20 mm by conventional techniques (e.g., physical exam for clinically palpable lymph nodes and superficial skin lesions or chest x-ray for clearly defined lung lesions surrounded by aerated lung) OR at least 10 mm by spiral CT scan or MRI
  * Nonmeasurable lesions, including the following:

    * Small lesions
    * Bone lesions
    * Pleural or pericardial effusions
    * Ascites
    * Irradiated lesions, unless progression is documented after radiotherapy
* Progressive or recurrent disease meeting at least 1 of the following criteria:

  * Measurable progressive disease
  * Biopsy-proven residual disease
  * Persistently elevated or rising ß-human chorionic gonadotropin (HCG) or alpha-fetoprotein (AFP) titers with no other clear cause for elevation
* Previously treated with 1 and only 1 regimen comprising etoposide and cisplatin with or without bleomycin AND exhibits clinical resistance by at least 1 of the following conditions after therapy*:

  * Progressive GCT after a partial response to first-line therapy
  * Relapse after complete response (CR) to first-line therapy, including partial response (PR) surgically converted to CR
  * Second testicular primary with evidence of metastases after first-line therapy
  * Relapse after adjuvant chemotherapy NOTE: *Patients failing to achieve PR or CR with first-line therapy as evidenced by rising markers or new disease within 4 weeks of first-line therapy are not eligible

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL (transfusion allowed)

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal* (ULN)
* AST and ALT ≤ 2.5 times ULN* NOTE: *Unless hepatic metastases are present

Renal

* Creatinine ≤ 1.5 times ULN OR
* Creatinine clearance ≥ 50 mL/min

Other

* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior dose-intensive therapy with stem cell replacement

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy
* No prior paclitaxel
* No prior docetaxel
* No prior ifosfamide
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy
* Concurrent or sequential radiotherapy to brain metastases allowed
* No other concurrent palliative radiotherapy

Surgery

* See Disease Characteristics
* Concurrent surgery for brain metastases allowed

Other

* Recovered from prior therapy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2004-04; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Motzer, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (79):
- United States (78):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Naval Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Palm Beach Cancer Institute - West Palm Beach, West Palm Beach, Florida
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at the Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., East Syracuse, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - NorthEast Oncology Associates - Concord, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Medical Center, Fayetteville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Comprehensive Cancer Center at Moore Regional Hospital, Pinehurst, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Miriam Hospital at Lifespan, Providence, Rhode Island
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Incorporated - Roanoke, Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
- McGill Cancer Centre at McGill University, Montreal, Quebec, Canada